CLINICAL TRIAL: NCT02465489
Title: Single-dose Pharmacokinetic Study of Deferiprone Extended Release Tablets Versus Ferriprox Immediate Release Tablets Under Fasting and Fed Conditions in Healthy Volunteers
Brief Title: Comparison of Deferiprone Extended Release Tablets and Ferriprox Immediate Release Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: LA51-0115
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: deferiprone; deferiprone extended release formulation; pharmacokinetics
MeSH Terms: interventions — Deferiprone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- ER, fasting conditions (Experimental): A single 1000 mg dose of deferiprone extended release tablet formulation administered under fasting conditions
  Interventions: Drug: Deferiprone extended release
- ER, fed conditions (Experimental): A single 1000 mg dose of deferiprone extended release tablet formulation administered under fed conditions
  Interventions: Drug: Deferiprone extended release
- ER half-tablets, fed conditions (Experimental): A single 1000 mg dose of deferiprone extended release tablet formulation (one 1000 mg tablet divided in two) administered under fed conditions
  Interventions: Drug: Deferiprone extended release
- IR, fasting conditions (Active Comparator): A single 1000 mg dose of deferiprone immediate release tablet formulation administered under fasting conditions
  Interventions: Drug: Deferiprone immediate release
- IR, fed conditions (Active Comparator): A single 1000 mg dose of deferiprone immediate release tablet formulation administered under fed conditions
  Interventions: Drug: Deferiprone immediate release

INTERVENTIONS:
Drug: Deferiprone extended release — Deferiprone 1000 mg extended release tablet formulation
  Other Names: Deferiprone extended release tablet formulation
  Arms: ER half-tablets, fed conditions; ER, fasting conditions; ER, fed conditions
Drug: Deferiprone immediate release — Ferriprox (deferiprone) 500 mg immediate release tablet formulation
  Other Names: Ferriprox immediate release tablet formulation
  Arms: IR, fasting conditions; IR, fed conditions

SUMMARY:
The purpose of this study is to look at the pharmacokinetics of a new formulation of deferiprone (deferiprone extended release tablets) under fed and fasting conditions.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, 5-period, 5-sequence study of the pharmacokinetics of a new formulation of deferiprone, extended release tablets, in twenty healthy volunteers. In each study period, blood samples for pharmacokinetics assessment will be collected pre-dose and over 24 hours post-dose. Safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 to <50 years
2. A female volunteer of childbearing potential must agree to use an accepted contraceptive regimen from at least 28 days prior to the first administration of the study drug until at least 30 days after the last dose of the study drug
3. A sexually active male must agree that he and/or his female partner will use a medically acceptable method of contraception throughout the study and for at least 30 days following drug administration
4. Body mass index (BMI) greater than or equal to 18.5 kg/m^2 and below 30.0 kg/m^2
5. Body weight of at least 60 kg
6. Non- or ex smoker
7. Clinical laboratory values within the laboratory's stated normal range; if not within this range, an abnormal value must be without any clinical significance
8. Have no clinically significant diseases captured in the medical history, or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, general biochemistry, coagulation, ECG, and urinalysis)

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Absolute neutrophil count (ANC) < 1.8 x 109/L at screening (no repeat can be performed)
3. History of significant hypersensitivity to deferiprone or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (such as angioedema) to any drugs
4. History or presence of gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs or known to potentiate or predispose to undesired effects
5. Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
6. Suicidal tendency, history of seizures, history of head trauma with coma or craniotomy/trepanation, state of confusion, or clinically relevant psychiatric diseases
7. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 220 msec, QRS < 60 msec, QRS >119 msec and QTcF > 450 msec for males and > 460 msec for females) on the screening ECG or other clinically significant ECG abnormalities
8. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
9. Any clinically significant illness in the previous 28 days before Day 1 of this study
10. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before Day 1 of this study
11. Any history of tuberculosis and/or prophylaxis for tuberculosis
12. Serum ferritin value below the normal limit of the reference laboratory at screening
13. Positive urine screening of alcohol and/or drugs of abuse
14. Positive results on HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAG (B) (hepatitis B)) or anti-Hepatitis C Virus (HCV (C)) tests
15. Positive result on a serum pregnancy test
16. Receipt of an investigational product in another clinical trial in the previous 28 days before Day 1 of this study
17. Donation of 50 mL or more of blood in the previous 28 days before Day 1 of this study or donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before Day 1 of this study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma Inc., Mount Royal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: Subjects were randomized to receive the following five treatments in different orders, with a 7-day washout period between treatments::
  A: Deferiprone ER tablets under fasting conditions B: Deferiprone ER tablets under fed conditions C: Deferiprone ER tablets administered as half-tablets under fed conditions D: Ferriprox IR tablets under fasting conditions E: Ferriprox IR tablets under fed conditions
  The sequences were as follows;
  * Sequence 1 (n=4): A-B-E-C-D
  * Sequence 2 (n=4): B-C-A-D-E
  * Sequence 3 (n=4): C-D-B-E-A
  * Sequence 4 (n=4): D-E-C-A-B
  * Sequence 5 (n=4): E-A-D-B-C
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 20
Completed | 15
Not Completed | 5
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteers: Subjects were randomized to receive five treatments in different orders:
  * deferiprone ER tablets under fasting conditions
  * deferiprone ER tablets under fed conditions
  * deferiprone ER tablets administered as half-tablets under fed conditions
  * Ferriprox IR tablets under fasting conditions
  * Ferriprox IR tablets under fed conditions
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  Canada | 20

OUTCOME MEASURES:

1. Primary Outcome: Cmax for Serum Deferiprone
Description: Maximum measured serum concentration. Blood samples will be collected pre-dose and over a 24-hour interval post-dose
Time Frame: Samples were collected pre-dose and at 0.25, 0.5, 0.75, 1.0, 1.33, 1.66, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 8.0, 12.0, 16.0, and 24.0 hours post-dose.
Population: The pharmacokinetic population included subjects who provided evaluable data for at least two study periods.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Extended Release, Fasting Conditions: A single 1000 mg dose of deferiprone extended release tablet formulation administered following a 10-hour fast
  Deferiprone extended release: Deferiprone 1000 mg extended release tablet formulation
- Extended Release, Fed Conditions: A single 1000 mg dose of deferiprone extended release tablet formulation administered following a high-fat breakfast
  Deferiprone extended release: Deferiprone 1000 mg extended release tablet formulation
- Extended Release Half-tablets, Fed Conditions: A single 1000 mg dose of deferiprone extended release tablet formulation (one 1000 mg tablet divided in two) administered following a high-fat breakfast
  Deferiprone extended release: Deferiprone 1000 mg extended release tablet formulation
- Immediate Release, Fasting Conditions: A single 1000 mg dose of Ferriprox immediate release tablet formulation administered following a 10-hour fast
  Deferiprone immediate release: Ferriprox (deferiprone) 500 mg immediate release tablet formulation
- Immediate Release, Fed Conditions: A single 1000 mg dose of Ferriprox immediate release tablet formulation administered following a high-fat breakfast
  Deferiprone immediate release: Ferriprox (deferiprone) 500 mg immediate release tablet formulation
Arm/Group | Extended Release, Fasting Conditions | Extended Release, Fed Conditions | Extended Release Half-tablets, Fed Conditions | Immediate Release, Fasting Conditions | Immediate Release, Fed Conditions
Number analyzed (Participants) | 16 | 16 | 14 | 16 | 15
μg/mL | 3.89 (1.47) | 2.76 (1.45) | 3.02 (1.03) | 13.89 (3.84) | 9.77 (3.60)

2. Primary Outcome: Tmax for Serum Deferiprone
Description: Time of maximum observed serum concentration. Blood samples will be collected pre-dose and over a 24-hour interval post-dose
Time Frame: as for outcome 1
Population: The pharmacokinetic population included subjects who provided evaluable data for at least two study periods
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Extended Release, Fasting Conditions | Extended Release, Fed Conditions | Extended Release Half-tablets, Fed Conditions | Immediate Release, Fasting Conditions | Immediate Release, Fed Conditions
Number analyzed (Participants) | 16 | 16 | 14 | 16 | 15
Hour | 3.63 (1.10) | 15.66 (9.33) | 8.29 (7.25) | 0.94 (0.63) | 1.91 (0.95)

3. Primary Outcome: AUC0-∞for Serum Deferiprone
Description: Area under the serum concentration time curve extrapolated to infinity. Blood samples will be collected pre-dose and over a 24-hour interval post-dose.
Time Frame: as for outcome 1
Population: The pharmacokinetic population included subjects who provided evaluable data for at least two study periods
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Extended Release, Fasting Conditions | Extended Release, Fed Conditions | Extended Release Half-tablets, Fed Conditions | Immediate Release, Fasting Conditions | Immediate Release, Fed Conditions
Number analyzed (Participants) | 15 | 2 | 5 | 16 | 15
ug*h/mL | 31.42 (6.68) | 40.52 (0.77) | 31.72 (8.21) | 34.81 (6.81) | 33.02 (7.19)

4. Secondary Outcome: Number of Subjects With Adverse Events (AEs)
Description: Number of subjects with AEs. AEs will include clinically significant changes from baseline in vital signs, 12-lead ECG, physical examinations, and laboratory tests.
Time Frame: Throughout the trial, from the time of the first dose until the last study visit (Day 36 or early termination)
Population: The safety population included all subjects who received at least one of the investigational products under study
Measure: Number; unit: participants
Arm/Group | Extended Release, Fasting Conditions | Extended Release, Fed Conditions | Extended Release Half-tablets, Fed Conditions | Immediate Release, Fasting Conditions | Immediate Release, Fed Conditions
Number analyzed (Participants) | 18 | 16 | 16 | 16 | 16
participants | 5 | 2 | 3 | 1 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the administration of the first dose in period 1 until the end-of-study visit
Arm/Group | Extended Release, Fasting Conditions | Extended Release, Fed Conditions | Extended Release Half-tablets, Fed Conditions | Immediate Release, Fasting Conditions | Immediate Release, Fed Conditions
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 5/18 | 2/16 | 3/16 | 1/16 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Release, Fasting Conditions (N=18) | Extended Release, Fed Conditions (N=16) | Extended Release Half-tablets, Fed Conditions (N=16) | Immediate Release, Fasting Conditions (N=16) | Immediate Release, Fed Conditions (N=16)
Amylase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Calcium Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Creatinine Increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Urine Present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-Reactive Protein Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural Dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine Odour Abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor retained title to and the right to publish all documentation, records, raw data, specimens or other work product generated in connection with the trial. Such publications shall not be made without the prior written consent of Sponsor. Neither Party will use the other Party's name in connection with any publication or promotion without the other Party's prior written consent. However, Sponsor has the right to publish appropriate information in order to satisfy regulatory requirements.